CLINICAL TRIAL: NCT02223559
Title: Non-invasive Assessment of Pulmonary Artery Pressure and Right Ventricular Function in Patients With Pulmonary Hypertension
Brief Title: Non-invasive Assessment of Pulmonary Artery Pressure
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Collaborators: National Bank of Austria (Other Government); Ludwig Boltzmann Institute for Lung Vascular Research (Other)
Responsible Party: Sponsor
Other Study IDs: 25-593 ex 12/13
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma samples will be retrained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- right heart catheterization patients

SUMMARY:
The assessment of pulmonary artery pressure (PAP) and parameters describing right ventricular function stand in the focus of the diagnosis and clinical management of pulmonary hypertension (PH). Right heart catheterization (RHC) is the gold standard method to measure PAP and to provide hemodynamic information on right ventricular function. However, due to its invasive nature, RHC is not optimal for screening and for close monitoring of the disease. Therefore, the development of non-invasive methods providing reliable PAP measurements and right ventricular functional parameters would be of major benefit.

Today, the most often used comprehensive non-invasive method for these purposes is echocardiography. However, the method has limitations; in many cases PAP is significantly under- or overestimated - especially in subjects with co-existing pulmonary diseases. Regarding right ventricular function, although novel echocardiography parameters appear to be promising, they have not yet been evaluated in all forms of PH.

Another emerging non-invasive method is cardiac magnetic resonance imaging (MRI). MRI is considered to be as gold standard for the non-invasive assessment of right ventricular function. In addition, our group showed that with a special approach ("vortex method"), MRI enables the determination of PAP with physiologic accuracy, but the method has not yet been validated systematically in different forms of PH.

All patients undergoing right heart catheterization in our clinic are candidates for the study. Excluded will be patients not eligible for MRI or declining to take part in the study. MRI and Echocardiography will be performed within two weeks of the RHC.

Hypothesis:

1. MRI is superior to echocardiography to non-invasively determine mean PAP in a broad collective of patients with PH of diverse ethology.
2. MRI derived right ventricular functional parameters correlate better to invasive measurements and to established prognostic parameters than echocardiography derived right ventricular functional parameters.
3. Novel right ventricular tissue Doppler parameters add substantially to "classical" echocardiography parameters to describe right ventricular function.

ELIGIBILITY:
Inclusion Criteria: patients undergoing right heart catheterization due to clinical reasons -

Exclusion Criteria: patients not eligible for MRI, patients not agreeing with investigation

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing right heart catheterization due to clinical reasons
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-08; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
mean pulmonary artery pressure | at baseline

SECONDARY OUTCOMES:
right ventricular function parameters | at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, Prof., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria